CLINICAL TRIAL: NCT02101736
Title: A Phase II Study of Cabozantinib (XL184) for Plexiform Neurofibromas in Subjects With Neurofibromatosis Type 1 in Children and Adults
Brief Title: Cabozantinib for Plexiform Neurofibromas (PN) in Subjects With NF1 in Children and Adults
Acronym: NF105-CABO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-130423015
Record Dates: First submitted 2014-03-14; First posted 2014-04-02 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: NF1; Neurofibromatosis; Plexiform Neurofibromas
Keywords: Cohort A: 3-15 years, Cohort B: Ages >= 16 years; Cabozantinib; XL184; Plexiform Neurofibromas; Neurofibromatosis; Pathogenetic NF1 Mutations; Cometriq; NF1
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma, Plexiform | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Cohort A: Single-arm open label two-stage Simon optimal study design Cohort B: Single-arm open-label study design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Agent XL184 (Cabozantinib) (Experimental): Cohort A (≥ 16 years - closed to accrual): Starting cabozantinib of 40 mg daily by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 60 mg based on dose tolerability. Subjects who do not tolerate 40 mg will dose reduce to 20 mg. Doses will be capped at 60 mg.
  Cohort B (3 - 15 years). The starting cabozantinib dose is 30 mg/m2/day by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 40 mg/m2/day based on dose tolerability. Subjects who do not tolerate 30 mg/m2/day will dose reduce to 23 mg/m2/day. Doses will be capped at 60 mg/day max daily dose
  Each cohort will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — This is an open label Phase II clinical trial. For both cohorts, subjects will receive cabozantinib orally in continuous cycles. Each cycle is 28 days. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with radiographic response (20% or greater reduction in tumor volume) at the end of 12 cycles can continue on therapy for up to an additional year. However, for Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study. For Cohort B, the criteria that subjects who do not achieve 15% reduction by 8 cycles are considered treatment failure and taken off study was eliminated. Subjects will be carefully monitored for toxicities associated with cabozantinib.
  Other Names: XL184; Cometriq

SUMMARY:
This study, "A Phase II Study of Cabozantinib (XL l84) for Plexiform Neurofibromas in Subjects with Neurofibromatosis Type I in Children and Adults diagnosed with Neurofibromatosis Type 1 (NF1) and have a type of tumor called a plexiform neurofibroma (PN). Neurofibromas are tumors that develop from the cells and tissues that cover the nerves. Plexiform neurofibromas can be disfiguring, painful, and life-threatening. These types of tumors typically do not respond well to most treatment approaches such as chemotherapy, radiation, and surgery because of their slow growth and location near vital structures of the body such as nerves, blood vessels, and the airway.

The primary objective is to determine the response rate of NF1 patients with plexiform neurofibromas treated with Cabozantinib therapy using MRI scans. The objective response rate to cabozantinib is defined as ≥ 20% reduction in tumor volume at the end of 12 cycles.

DETAILED DESCRIPTION:
There are two cohorts: Cohort A is for patients ≥ 16 years of age and Cohort B is for patients 3 - 15 years of age. Cohort A is closed to enrollment but this study will open to Cohort B patients. This phase II open label study will evaluate adults and children with NF1 and plexiform neurofibromas treated with cabozantinib (XL184). This study will enroll subjects who either meet clinical diagnostic criteria or have an identified pathogenetic NF1 mutation. Subjects on study must have clinically significant plexiform neurofibroma defined as potentially life-threatening, impinging on vital structures or significantly impairing the quality of life from pain or other symptoms. Patients must not have lesions suspicious for malignant tumors such as MPNSTs (malignant peripheral nerve sheath tumors) and suspicious tumors must be proven negative by histopathology prior to enrollment on study. Since Cohort A is closed to accrual, this study will be open to Cohort B, patients 3 - 15 years of age that meet eligibility criteria.

For Cohort A, the study will be a Simon two-stage study design. It will be a single-arm open-label study of cabozantinib and the primary endpoint is the objective response rate (ORR) to cabozantinib at 1 year. In the first stage, 9 evaluable subjects will be accrued. If there is at least 1 response, accrual will continue to the second stage and an additional 8 evaluable subjects will be enrolled. To allow for 25% unevaluable subjects, a maximum of 24 subjects will be enrolled. Radiographic response will be evaluated as the primary endpoint with 20% volumetric MRI response of the target lesion being the threshold criteria for tumor response. A target lesion will be selected at time of enrollment and tumor evaluations will occur serially while on study.

For Cohort B, a minimum of 17 evaluable subjects will be enrolled. To allow for up to 25% unevaluable subjects, a minimum of 24 subjects will be enrolled. Based on preliminary response data and minimal toxicity in Cohort A, a 2-stage design is not felt to be necessary for Cohort B.

In Cohort A, all subjects will start cabozantinib at 40 mg. The published maximum tolerated dose (MTD) for Cabozantinib is 140 mg and the current recommended dose in Phase 3 clinical trials for subjects with medullary thyroid cancer is 100 mg. Doses of 40 mg and 60 mg continue to show efficacy in on-going phase 2 and phase 3 trials with reduced toxicity. Subjects who tolerate 40 mg for 2 cycles will escalate to 60 mg. The rationale for this is that the majority of subjects who develop toxicity do so after >2 weeks on drug as cabozantinib has a long half-life. Subjects who experience dose-limiting toxicity at 40 mg will dose reduce to 20 mg when their toxicities resolve. Subjects without toxicity at 40mg will increase to 60mg. Subjects who experience toxicity at 60 mg will dose reduce to 40 mg. This dosing schema is designed to maximize safety and tolerability in this new population of patients.

In Cohort B, subjects will start at 30 mg/m2/day dosing. Dose will be escalated at cycle 3 if tolerated to 40 mg/m2. Subjects who experience DLT at 40 mg/m2/day will dose reduce to 30 mg/m2/day. Subjects who experience DLT at 30 mg/m2/day will dose reduce to 23 mg/m2day. Actual dosing will be based on the dosing nomogram.

Dosing will be continuous, with 28 days defined as a cycle and each cycle reporting period is day 1 to day 28. In the absence of progressive disease or dose limiting toxicity (DLT), subjects may continue on therapy for a total of 12 total cycles. Subjects who have a radiographic response (20% or greater reduction in tumor volume) on therapy at the end of 12 cycles can continue on therapy for up to an additional year. The maximum duration for treatment under this study design is 24 cycles. However, subjects who do not achieve at least 15% reduction in index tumor volume after 8 cycles (~8 months) will be considered treatment failures and taken off study. Subjects entered on the trial will be carefully monitored for the development of cabozantinib associated toxicities, and target modifications and interruptions will be performed.

The investigational nature and objectives of this trial, the procedures and treatment involved, the risks, discomforts, and benefits, and potential alternatives therapies will be carefully explained to the subject and/or subject's parent(s) or guardian, if subject is a child,by the site Principal Investigator or designated associate investigator. When appropriate, pediatric patients will be included in all discussions. A signed informed consent document will be obtained prior to determining eligibility and entry criteria to this trial. Subjects entered on this trial will be treated with therapeutic intent and response to therapy will be closely monitored. This protocol involves greater than minimal risk but presents the potential for direct benefit to individual subjects

Schedule of study evaluations are summarized below:

Pre-Study:

* Medical history, physical exam with vital signs, blood pressure, and pulse oximetry
* Performance status to assess your ability to perform everyday tasks
* Laboratory tests including blood and urine tests for routine safety tests
* Urine pregnancy test for females of childbearing age
* Electrocardiogram (EKG) to monitor the electrical activity of the heart
* MRI of neurofibromas
* Completion of health-related questionnaires on quality of life, pain assessment, and PN symptom checklist (upon study entry)
* Research blood draws ( 2 tablespoons) to evaluate the tumor's response to treatment and the action of cabozantinib in the body over a period of time (Upon study entry on Cycle 1 Day 1, predose and 4-hours post dose)

During Study Treatment:

End of Cycles 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, 18, 20, 22, 24 or Early Termination (additional visit that is not within the specified times mentioned.)

* Medical History
* Physical exam with vital signs, blood pressure and pulse oximetry
* Performance Status
* Review of Subject Diary
* Urine pregnancy test for females of childbearing age at end of cycles 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
* Electrocardiogram (EKG) to monitor the electrical activity of the heart at end of cycles 1, 2, 4, 6, 9, 12, 16, 20, 24

End of Cycles 1 - 24, or Early Termination

* Laboratory tests including blood and urine tests for routine safety tests

End of Cycles 4, 8, 12, 18, 24, or Early Termination

* MRI of neurofibromas
* Completion of health-related questionnaires on quality of life, pain assessment, and PN symptom checklist

Cycles 1, 2, 3, 4

* Research blood draws ( 2 tablespoons) to evaluate the tumor's response to treatment and the action of cabozantinib in the body over a period of time

Phone Calls will be made at the end of cycles 13, 15, 17, 19, 21, and 23 to assess drug compliance and toxicity

The protocol PI and clinical coordinator will review the subject eligibility, study progress, safety issues, protocol deviations and adverse events. A Data Safety Monitoring Board (DSMB) and a medical monitor has been established for the purpose of ensuring data compliance and regular monitoring of this trial. The medical monitor is a qualified physician and is not associated with this particular protocol. The medical monitor is specifically required to review all unanticipated problems involving risk to subjects or others, serious adverse events and deaths associated with the protocol and provide an unbiased written report of the event.

An early stopping rule will be invoked for both cohorts to potentially prevent accrual of subjects onto the study in the event that Cabozantinib is associated with a higher than acceptable rate of dose-limiting toxicity (DLT) requiring removal from study (set at 10% or higher) during the first 2 cycles. Toxicity will be continuously monitored. If at any time >2 of the first 10 subjects or 4 or more of the first 15 total subjects are removed for DLT, then accrual will be stopped until the DSMB reviews safety and efficacy data for the study and recommends termination or despite the DLT (because of the benefit:risk assessment or other reasoning) recommends reopening recruitment. Boundaries for DSMB for consideration of terminating each cohort (both cohort A and B) would be the same.

The sample size for this trial is based on the safety and feasibility factors. The data needed is based on risk versus benefit. For feasibility, we expect at least efficacy of a 25% response rate. For safety reasons, subjects who do not achieve at least a 15% reduction in tumor volume will not be continued beyond 8 courses, as the likelihood of achieving a response (20% reduction in tumor volume) by 12 months is minimal. These subjects will be discontinued from the trial and counted in an "Intent to Treat" analysis as evaluable and as failures.

All analyses for outcome results will be based on evaluable subjects. Definitions of evaluable include: 1.) Evaluation for toxicity (subject who received at least one dose of study drug and removed from treatment for toxicity are evaluable. Any subject who completed one full cycle of therapy is evaluable for toxicity); 2.)Evaluation for response (subjects who have completed at least two cycles of therapy and have had their first follow-up MRI evaluation. Subjects who did not respond and are later found to have a target tumor other than a plexiform neurofibroma (e.g. malignant peripheral nerve sheath tumor) are not evaluable for response).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or molecular diagnosis of Neurofibromatosis Type 1
2. Plexiform neurofibroma that is progressive OR causing significant morbidity.
3. Measurable disease amenable to volumetric MRI imaging defined as lesion seen on at least 3 consecutive MRI slices and at least 3 mL in volume. Select tumors <3 cm may be eligible on review.
4. Central review or MRI required prior to enrollment.
5. Age ≥ 3 years of age at the time of study entry. Subjects ≥ 16 years will be enrolled in Cohort A. Subjects 3 - 15 years will be enrolled in Cohort B.
6. Performance Level Karnofsky ≥ 50%. Subjects unable to walk because of paralysis, but up in a wheel chair will be considered ambulatory for purpose of assessing performance score.
7. Complete resection of plexiform neurofibroma is not feasible or if subject refuses surgery.
8. Fully recovered from acute toxic effects of all prior chemotherapy or radiotherapy.
9. No myelosuppressive chemotherapy within 4 weeks of study entry.
10. At least 7 days since completion of hematopoietic growth factors.
11. At least 14 days since completion of biologic agent.
12. At least 4 weeks since receiving any investigational drug.
13. Physiologic or stress doses of steroids allowed in patients with endocrine deficiencies.
14. At least 6 months from radiation therapy to index tumor and at least 6 weeks from radiation to areas outside of index plexiform neurofibroma.
15. At least 3 months from major surgery or at least 1 month from minor surgery. No major surgery anticipated within 3 months of enrollment.
16. Adequate bone marrow function.
17. Adequate renal function.
18. Adequate liver function.
19. Blood pressure within upper limit of normal.

Exclusion Criteria:

1. Active optic glioma or other low-grade glioma requiring treatment with chemotherapy or radiation therapy.
2. Malignant glioma, malignant peripheral nerve sheath tumor, or other malignancy requiring treatment in the last 12 months.
3. Dental braces or prosthesis that interferes with volumetric analysis of the neurofibroma(s).
4. Unable to swallow tablets.
5. Women who are pregnant or breast-feeding.
6. Subjects of reproductive potential who have not agreed to use effective contraception.
7. Subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs).
8. Subject requires anticoagulants. Low dose aspirin, low-dose warfarin, and prophylactic low molecular weight heparin are permitted.
9. Concomitant treatment of strong CYP3A4 inducers or inhibitors.
10. History of noncompliance to medical regimens
11. A known history of HIV seropositivity or known immunodeficiency. HIV testing will not be required as part of this trial, unless HIV is clinically suspected.
12. Impairment of gastrointestinal function or gastrointestinal disease that may affect the absorption of cabozantinib. (e.g. ulcerative disease, malabsorption syndrome, or small bowel resection). Nasogastric tube (NG) tube is allowed.

    * Any of the following within 28 days before the first dose of study treatment:

      1. intra-abdominal tumor/metastases invading GI mucosa
      2. active peptic ulcer disease
      3. inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      4. malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      1. abdominal fistula
      2. gastrointestinal perforation
      3. bowel obstruction or gastric outlet obstruction
      4. intra-abdominal abscess. Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating study treatment even if abscess occurred more than 6 months before the first dose of study treatment.
    * Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
13. Patients who have an uncontrolled infection.
14. Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
15. Hemoptysis of ≥0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
16. Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
17. Radiographic evidence of cavitating pulmonary lesion(s).
18. Concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration)
19. Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days before the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Baseline heart-rate corrected QT (QTc) interval >470 msec in women and >450 msec in men
    * Concomitant treatment with medications that prolong the QT interval and have a known risk of Torsades de Pointes is not contraindicated, but should be avoided if possible and will require more frequent EKG monitoring.
    * Any of the following within 6 months before the first dose of study treatment:

      1. unstable angina pectoris
      2. clinically-significant cardiac arrhythmias
      3. stroke (including transient ischemic attack (TIA), or other ischemic event)
      4. myocardial infarction
      5. thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
20. Other clinically significant disorders such as:

    * Active infection requiring systematic treatment within 28 days before the first dose of study treatment
    * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
    * History of organ transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
21. Complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of study treatment irrespective of time from surgery.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chie-Schin Shih, MD, Principal Investigator — Indiana University
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana Unversity, Indianapolis, Indiana
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Children' Hospital Boston and Massachusetts General Hospital, Boston, Massachusetts
  - Washington University - St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Fisher MJ, Shih CS, Rhodes SD, Armstrong AE, Wolters PL, Dombi E, Zhang C, Angus SP, Johnson GL, Packer RJ, Allen JC, Ullrich NJ, Goldman S, Gutmann DH, Plotkin SR, Rosser T, Robertson KA, Widemann BC, Smith AE, Bessler WK, He Y, Park SJ, Mund JA, Jiang L, Bijangi-Vishehsaraei K, Robinson CT, Cutter GR, Korf BR; Neurofibromatosis Clinical Trials Consortium; Blakeley JO, Clapp DW. Cabozantinib for neurofibromatosis type 1-related plexiform neurofibromas: a phase 2 trial. Nat Med. 2021 Jan;27(1):165-173. doi: 10.1038/s41591-020-01193-6. Epub 2021 Jan 13. PMID 33442015
- [Derived] Armstrong AE, Brossier NM, Hirbe AC. Neurofibromatosis type 1-related tumours in paediatrics: an evolving treatment landscape. Lancet Child Adolesc Health. 2020 Jul;4(7):488-490. doi: 10.1016/S2352-4642(20)30169-3. No abstract available. PMID 32562630

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with 20% or greater reduction in tumor volume at the end of 12 cycles can continue on therapy for up to an additional year. However, for Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study. For Cohort B, the criteria that subjects who do not achieve 15% reduction by 8 cycles are considered treatment failure and taken off study was eliminated.
Groups:
- Cohort A: Cohort A (≥ 16 years - closed to accrual): Starting cabozantinib of 40 mg daily by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 60 mg based on dose tolerability. Subjects who do not tolerate 40 mg will dose reduce to 20 mg. Doses will be capped at 60 mg.
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. Subjects will receive cabozantinib orally in continuous 28 day cycles. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with 20% or greater reduction in tumor volume at the end of 12 cycles can continue on therapy for up to an additional year. However, for Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study.
- Cohort B: Cohort B (3 - 15 years). The starting cabozantinib dose is 30 mg/m2/day by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 40 mg/m2/day based on dose tolerability. Subjects who do not tolerate 30 mg/m2/day will dose reduce to 23 mg/m2/day. Doses will be capped at 60 mg/day max daily dose.
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. Subjects will receive cabozantinib orally in continuous 28 day cycles. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with 20% or greater reduction in tumor volume at the end of 12 cycles can continue on therapy for up to an additional year. For Cohort B, the criteria that subjects who do not achieve 15% reduction by 8 cycles are considered treatment failure and taken off study was eliminated.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 23 | 22
Completed | 19 | 21
Not Completed | 4 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: Cohort A (≥ 16 years - closed to accrual): Starting cabozantinib of 40 mg daily by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 60 mg based on dose tolerability. Subjects who do not tolerate 40 mg will dose reduce to 20 mg. Doses will be capped at 60 mg.
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. Subjects will receive cabozantinib orally in continuous 28 day cycles. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with 20% or greater reduction in tumor volume at the end of 12 cycles can continue on therapy for up to an additional year. For Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study.
- Cohort B: Cohort B (3 - 15 years). The starting cabozantinib dose is 30 mg/m2/day by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 40 mg/m2/day based on dose tolerability. Subjects who do not tolerate 30 mg/m2/day will dose reduce to 23 mg/m2/day. Doses will be capped at 60 mg/day max daily dose
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. Subjects will receive cabozantinib orally in continuous 28 day cycles. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with 20% or greater reduction in tumor volume at the end of 12 cycles can continue on therapy for up to an additional year. For Cohort B, the criteria that subjects who do not achieve 15% reduction by 8 cycles are considered treatment failure and taken off study was eliminated.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There are two cohorts. Cohort A had 23 subjects at baseline and Cohort B had 22 subjects at baseline. The overall total was 45 subjects at baseline.
  years | 23.3 (5.49) | 10 (4.28) | 16.65 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are two cohorts. Cohort A had 23 subjects at baseline and Cohort B had 22 subjects at baseline. The overall total was 45 subjects at baseline.
  Participants
    Female | 9 | 11 | 20
    Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are two cohorts. Cohort A had 23 subjects at baseline and Cohort B had 22 subjects at baseline. The overall total was 45 subjects at baseline.
  Participants
    Hispanic or Latino | 0 | 3 | 3
    Not Hispanic or Latino | 22 | 19 | 41
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are two cohorts. Cohort A had 23 subjects at baseline and Cohort B had 22 subjects at baseline. The overall total was 45 subjects at baseline.
  Participants
    Overall Study: American Indian or Alaska Native | 0 | 0 | 0
    Overall Study: Asian | 2 | 1 | 3
    Overall Study: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Overall Study: Black or African American | 1 | 3 | 4
    Overall Study: White | 17 | 16 | 33
    Overall Study: More than one race | 0 | 0 | 0
    Overall Study: Unknown or Not Reported | 2 | 2 | 4
Volumetric Response [Median (Full Range); unit: mm^3] — Evaluable subjects for tumor volume in mm^^3 Population: There are two cohorts with different numbers of evaluable subjects in each.
  mm^3
    number analyzed (Participants) | 19 | 21 | 40
    (all) | 556.6 [56.8 to 2954] | 355.1 [32.9 to 4068.7] | 455.9 [56.8 to 4068.7]

OUTCOME MEASURES:

1. Primary Outcome: The Change in Tumor Size Based on Radiographic Assessment
Description: We will estimate the objective response rate (ORR) as defined by 20% volumetric MRI response of the target lesion to cabozantinib at 12 months in adolescents and adults with Neurofibromatosis type 1 (NF1) plexiform neurofibromas by volumetric MRI imaging.
Time Frame: baseline to 12 Months
Population: There were a total of 19 evaluable subjects from Cohort A and 21 for Cohort B.
Measure: Median (Full Range); unit: mm^3
Groups:
- Cohort A: Cohort A (≥ 16 years - closed to accrual): Starting cabozantinib of 40 mg daily by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 60 mg based on dose tolerability. Subjects who do not tolerate 40 mg will dose reduce to 20 mg. Doses will be capped at 60 mg.
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. For both cohorts, subjects will receive cabozantinib orally in continuous cycles. Each cycle is 28 days. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with radiographic response (20% or greater reduction in tumor volume) at the end of 12 cycles can continue on therapy for up to an additional year. For Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study.
- Cohort B: Cohort B (3 - 15 years). The starting cabozantinib dose is 30 mg/m2/day by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 40 mg/m2/day based on dose tolerability. Subjects who do not tolerate 30 mg/m2/day will dose reduce to 23 mg/m2/day. Doses will be capped at 60 mg/day max daily dose
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. For both cohorts, subjects will receive cabozantinib orally in continuous cycles. Each cycle is 28 days. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with radiographic response (20% or greater reduction in tumor volume) at the end of 12 cycles can continue on therapy for up to an additional year. For Cohort B, the criteria that subjects who do not achieve 15% reduction by 8 cycles was eliminated.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 19 | 21
mm^3 | -15.7 [-38 to 2.8] | -4.1 [-25.8 to 12.5]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: This is the number of participants with one or more adverse events.
Time Frame: baseline to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Cohort A (≥ 16 years - closed to accrual): Starting cabozantinib of 40 mg daily by mouth per cycle. Duration of each cycle is 28 days. Subjects will dose escalate after 2 cycles to 60 mg based on dose tolerability. Subjects who do not tolerate 40 mg will dose reduce to 20 mg. Doses will be capped at 60 mg.
  Each cohort A and B will enroll up to 24 evaluable subjects with a target minimum of 17 evaluable subjects per cohort.
  Cabozantinib: This is an open label Phase II clinical trial. For both cohorts, subjects will receive cabozantinib orally in continuous cycles. Each cycle is 28 days. In absence of progressive disease or dose limiting toxicity (DLT), subjects may continue therapy for a total of 24 cycles. Subjects with radiographic response (20% or greater reduction in tumor volume) at the end of 12 cycles can continue on therapy for up to an additional year. However, for Cohort A, subjects who do not achieve 15% reduction in tumor volume after 8 cycles will be considered treatment failure and taken off study.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 23 | 22
Participants | 20 | 21

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of dose (baseline) up to 2 years.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/23 | 5/22
Other Adverse Events (participants affected / at risk) | 21/23 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=23) | Cohort B (N=22)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
SKIN INFECTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABSCESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIFFICULTY WALKING, BACK PAIN, BOWEL/BLADDER URGENCY, LEGS GAVE OUT, AND PARESTHESIAS (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
SUBJECT WAS ADMITTED TO THE HOSPITAL ON 10/24/20 WITH GRADE 2 WEIGHT LOSS THAT THE PHYSICIAN FELT NE (Investigations) | 0 (0) | 1 (1)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=23) | Cohort B (N=22)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (2) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 2 (6) | 1 (2)
VERTIGO (Ear and labyrinth disorders) | 2 (4) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 1 (2) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 4 (5) | 21 (32)
BLURRED VISION (Eye disorders) | 9 (38) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (7) | 6 (9)
BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (8) | 3 (4)
DIARRHEA (Gastrointestinal disorders) | 3 (8) | 16 (33)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 2 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 9 (17)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 2 (4) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (4) | 9 (20)
FATIGUE (General disorders) | 1 (1) | 11 (18)
PAIN (General disorders) | 1 (1) | 7 (15)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (5) | 8 (11)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 17 (101) | 0 (0)
PARONYCHIA (Infections and infestations) | 3 (13) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ABSOLUTE LYMPHOCYTE COUNT INCREASED (Investigations) | 1 (1) | 0 (0)
ABSOLUTE NEUTROPHIL COUNT DECREASED (Investigations) | 4 (6) | 2 (3)
ABSOLUTE NEUTROPHIL COUNT INCREASED (Investigations) | 13 (38) | 0 (0)
ALANINE AMINOTRANSFERASE DECREASED (Investigations) | 3 (5) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 9 (12)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (2) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 9 (18)
BILIRUBIN INCREASED (Investigations) | 3 (8) | 3 (6)
BUN INCREASED (Investigations) | 10 (55) | 0 (0)
HEMOGLOBIN INCREASED (Investigations) | 1 (6) | 4 (4)
LIPASE INCREASED (Investigations) | 1 (1) | 2 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (2) | 2 (3)
PLATELET COUNT DECREASE (Investigations) | 1 (1) | 5 (5)
SERUM AMYLASE INCREASED (Investigations) | 1 (1) | 1 (1)
SKIN INFECTION (Infections and infestations) | 6 (8) | 1 (1)
THYROID STIMULATING HORMONE INCREASED (Endocrine disorders) | 1 (1) | 0 (0)
WEIGHT GAIN (Investigations) | 4 (8) | 2 (6)
WEIGHT LOSS (Investigations) | 18 (32) | 12 (21)
WHITE BLOOD CELL INCREASED (Investigations) | 3 (4) | 0 (0)
ANOREXIA (Investigations) | 2 (3) | 9 (13)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (8) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (20) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (3) | 2 (5)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (2) | 4 (8)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3 (8) | 1 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (6) | 5 (8)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (2) | 4 (7)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (2) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 6 (6) | 0 (0)
HEADACHE (Nervous system disorders) | 10 (55) | 8 (9)
ANXIETY (Psychiatric disorders) | 1 (3) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 6 (26) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 3 (4) | 7 (9)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (3) | 0 (0)
URINARY URGENCY (Renal and urinary disorders) | 3 (7) | 1 (1)
IRREGULAR MENSTRUATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
ACNEIFORM RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CALLUS OF FOOT (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
HAIR COLOR CHANGE (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (5)
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
MACULOPAPULAR RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (17)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
TINEA PEDIS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
FLUSHING (Vascular disorders) | 6 (23) | 0 (0)
HOT FLASHES (Vascular disorders) | 9 (26) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (2) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3) | 4 (4)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Behaviour Disturbance (Psychiatric disorders) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 10 (55) | 3 (6)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 9 (21) | 0 (0)
Cold Sore (Infections and infestations) | 4 (7) | 0 (0)
Concentration Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 0 (0) | 2 (7)
Decreased Platelet Count (Investigations) | 3 (10) | 5 (5)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0)
Ear And Labyrinth Disorders - Other, Impacted Cerumen (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Elevated Amylase (Investigations) | 0 (0) | 1 (1)
Emotional Lability (Psychiatric disorders) | 5 (18) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Disorders - Other, Buccal Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorders - Other, Dental Pain (Gastrointestinal disorders) | 2 (4) | 1 (1)
Gastrointestinal Disorders - Other, Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 4 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infections And Infestations - Other, Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Infections And Infestations - Other, Gi Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Injury, Poisoning And Procedural Complications - Other, Ankle Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, Poisoning And Procedural Complications- Other, Scalp Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigations - Other, Eosinophilia (Investigations) | 1 (1) | 1 (1)
Investigations - Other, Increased Mean Corpuscular Volume (Investigations) | 0 (0) | 1 (1)
Investigations - Other, International Normalized Ration Increased (Investigations) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 15 (82) | 0 (0)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Localized Edema (General disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (2)
Metabolism And Nutrition Disorders - Other, Decreased Oral Intake (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism Other - Decreased Vitamin D (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metbolism And Nutrition Disorders - Other, Hyperchloremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (2)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 4 (22) | 1 (1)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal And Connective Tissue Disorder - Other, Tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal And Connective Tissue Disorders - Other, Extremity Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (11) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 5 (7) | 9 (20)
Pale Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 8 (24) | 0 (0)
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (2) | 1 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Platelet Count Decreased (Investigations) | 1 (1) | 5 (5)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Psychiatric Disorders - Other, Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
Rash Ezcematoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Renal & Urinary Disorders - Other, Ketonuria (Renal and urinary disorders) | 0 (0) | 5 (7)
Scalp Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (6) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin And Subcutaneous Disorders - Other, Achromotricia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin And Subcutaneous Disorders - Other, Dry Skin Patches (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin And Subcutaneous Tissue Disorders - Other, Skin Color Change (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin And Subcutaneous Tissue Disorders - Other: Blue Lips (Not Cyanosis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin And Subcutaneous Tissue Disorders- Other, Blister/Bug Bite On Finger (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin And Subcutaneous Tissue Disorders- Other, Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Skin And Subcutaneous Tissue Disorders- Other, New Freckles/Moles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin And Subcutaneous Tissue Disorders- Other, Rash Unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Skin And Subcutaneous Tissue Disorders- Other, Sore On Lips (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3)
Skin And Subcutaneous Tissue Disorders- Other, Transient Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Blisters (Skin and subcutaneous tissue disorders) | 10 (50) | 0 (0)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Surgical & Medical Procedures - Other, Dental Extractions (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (7) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 6 (22) | 0 (0)
Total Protein Level Increased (Investigations) | 8 (34) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 4 (8)
Urine Discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine White Blood Cell Increased (Investigations) | 2 (6) | 0 (0)
Urobilinogen Increased (Investigations) | 4 (7) | 0 (0)
Vitamin D Deficiency (Immune system disorders) | 3 (5) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 15 (28) | 6 (7)
White Blood Cell Count Increased (Investigations) | 2 (7) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02101736/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT02101736/ICF_001.pdf